CLINICAL TRIAL: NCT07001787
Title: A Phase I, Randomized, Double-Blind, Placebo-controlled Study to Assess the Safety, Tolerability，Pharmacokinetics, and Pharmacodynamics of HS-10510 Following Single and Multiple Ascending Dose Administration to Healthy Subjects With or Without Elevated LDL-C Levels
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HS-10510 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-10510-101
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Dyslipidemia
Keywords: Elevated LDL-C；Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part A-HS-10510 dose 1/placebo (Active Comparator): A total of 6 subjects will receive single ascending doses of HS-10510 and 2 will receive placebo
  Interventions: Drug: Drug：HS-10510；; Drug: Drug：Placebo
- Part A-HS-10510 dose 2/placebo (Active Comparator): A total of 6 subjects will receive single ascending doses of HS-10510 and 2 will receive placebo
  Interventions: Drug: Drug：HS-10510；; Drug: Drug：Placebo
- Part A-S-10510 dose 3/placebo (Active Comparator): A total of 6 subjects will receive single ascending doses of HS-10510 and 2 will receive placebo
  Interventions: Drug: Drug：HS-10510；; Drug: Drug：Placebo
- Part A-HS-10510 dose 4/placebo (Active Comparator): A total of 6 subjects will receive single ascending doses of HS-10510 and 2 will receive placebo
  Interventions: Drug: Drug：HS-10510；; Drug: Drug：Placebo
- Part B-HS-10510 dose 1/placebo (Active Comparator): A total of 9 subjects will receive multiple ascending doses of HS-10510 and 3 will receive placebo
  Interventions: Drug: Drug：HS-10510；; Drug: Drug：Placebo
- Part B-HS-10510 dose 2/placebo (Active Comparator): A total of 9 subjects will receive multiple ascending doses of HS-10510 and 3 will receive placebo
  Interventions: Drug: Drug：HS-10510；; Drug: Drug：Placebo
- Part B-HS-10510 dose 3/placebo (Active Comparator): A total of 9 subjects will receive multiple ascending doses of HS-10510 and 3 will receive placebo
  Interventions: Drug: Drug：HS-10510；; Drug: Drug：Placebo
- Part C-HS-10510/Placebo with rosuvastatin (Active Comparator): A total of 10 subjects will receive HS-10510 in combination with rosuvastatin and 10 subjects will receive placebo in combination with rosuvastatin
  Interventions: Drug: Drug：HS-10510；; Drug: Drug：Placebo; Drug: Drug： Rosuvastatin

INTERVENTIONS:
Drug: Drug：HS-10510； — Drug：HS-10510 Description：Subjects will receive HS-10510 orally as a single and multiple ascending dose.
Drug: Drug：Placebo — Drug：Placebo Description：Subjects will receive placebo matching the HS-10510 dose orally as a single and multiple ascending dose.
Drug: Drug： Rosuvastatin — Drug：Rosuvastatin Description：Subjects will receive rosuvastatin orally.
  Arms: Part C-HS-10510/Placebo with rosuvastatin

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of HS-10510 following single and multiple dose administration to healthy subjects with or without elevated Low-Density Lipoprotein-Cholesterol (LDL-C) levels.

This study will consist of three parts (Parts A，B and C). 32 subjects have been planned for Part A and up to 36 subjects for Part B and 20 subjects for Part C.

DETAILED DESCRIPTION:
This is a Phase I, First In Human (FIH), randomized, double-blind, placebo-controlled, study in Chinese healthy male and female subjects at one center. 32 subjects have been planned for Part A and up to 36 subjects for Part B and 20 subjects for Part C.

* Part A（SAD cohort）: A Screening Period of maximum 28 days. Admission to study center (Day -1). A Treatment Period (Day 1 to Day 4) with a single dose of HS-10510 or placebo on Day 1. Subjects will be discharged on Day 4. A Follow-up Visit within 7 days after the Investigational Medicinal Product (IMP) dose for all cohorts. (i) Part A1 - Up to 4 dose cohorts of HS-10510 are planned to be investigated. Within each cohort, 6 subjects will be randomized to receive HS-10510, and 2 subjects randomized to receive placebo. (ii) Part A2 - The subjects from a chosen cohort in Part A1 will stay at study center for 7 days to wash out after the first dose administration of IMP and will receive HS-10510 or placebo after intake of a high-calorie, high-fat breakfast, to assess the effect of food on the PK of HS-10510. The subjects will stay at the study center until 72 hours post-dose in both the parts.
* Part B（MAD cohort）: Up to 3 dose cohorts are planned to be investigated. In each cohort, 12 subjects will participate and receive either HS-10510 or placebo, randomized 3:1 for 28 days dosing.
* Part C（Rosuvastatin MAD cohorts）：20 subjects in this cohort will receive either HS-10510 in combination with rosuvastatin (10 subjects) or placebo in combination with rosuvastatin (10 subjects). Subjects eligible for these cohorts will begin a Screening period of 28 days, a rosuvastatin run-in period of 28 days, Treatment period of 28 days for this cohort and one Follow-up visits (1 week after last dose of IMP).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged 18-55 years (inclusive) at the time of signing the informed consent form.
2. Agree to use highly effective contraception from the date of signing the informed consent to 30 days after the last dose.
3. Male or female subjects agree to avoid donating sperm or eggs from the date of signing the informed consent to 90 days after the last dose.
4. Female subjects of childbearing potential must have a negative blood pregnancy test within 3 days before dosing.
5. Based on the medical history, physical examination, vital signs (VS) measurements, and ECG and safety test results conducted during the screening visit and before randomization, the subject is in good health.
6. The subject has a full understanding of the trial content, process, and potential adverse reactions, is willing to strictly adhere to the trial protocol to complete this study, and voluntarily signs the informed consent form.
7. No more than 14 units of alcohol (1 unit = 285 mL of beer, 25 mL of spirits, 125 mL of wine) in a single session within two weeks before screening; no alcohol (including alcohol-containing products) 48 hours before dosing and throughout the study period.
8. No smoking 48 hours before dosing and throughout the study period.
9. No more than 6 cups (approximately 250 mL per cup) of coffee, tea, cola, or other caffeine-containing beverages on average per day within three months before screening; no xanthine- or caffeine-containing foods or beverages throughout the study period.
10. Maintain a stable diet and exercise lifestyle throughout the study period; avoid all activities that may cause injury or intense physical activity.
11. Agree to avoid consuming grapefruit, grapefruit juice, bitter orange, bitter orange juice, or other products containing grapefruit or bitter orange, mulberry juice, cruciferous vegetables (such as kale, watercress, Chinese broccoli, Brussels sprouts, and mustard greens), or grilled meats from 7 days before dosing to the end of the last visit.

    For Part A
12. BMI between 19.0-28.0 kg/m2 (inclusive), with a minimum weight of 50.0 kg for males and 45.0 kg for females.

    For Part B
13. Fasting LDL-C between 1.8-4.9 mmol/L (inclusive) at screening.
14. Fasting triglycerides ≤4.52 mmol/L at screening.
15. BMI between 20.0-35.0 kg/m2 (inclusive), with a minimum weight of 50.0 kg for males and 45.0 kg for females.

    For Part C
16. Fasting LDL-C between 2.6-4.9 mmol/L (inclusive) at screening.
17. Fasting triglycerides ≤4.52 mmol/L at screening.
18. BMI between 20.0-35.0 kg/m2 (inclusive), with a minimum weight of 50.0 kg for males and 45.0 kg for females.
19. LDL-C reduction of ≥30% after a 28-day rosuvastatin run-in period.

Exclusion Criteria:

1. Subjects with clinically significant abnormalities in vital signs, physical examination, or laboratory test results during the screening period, as determined by the investigator (a single retest may be performed within the screening window if there is a clear reason for retesting, and the retest results will be used for screening).
2. Subjects who have undergone LDL apheresis or plasmapheresis within 12 months before screening.
3. Subjects who have donated or lost ≥400 mL of blood or received a blood transfusion or bone marrow donation within 3 months before screening; or donated or lost ≥200 mL of blood within 1 month before screening.
4. Subjects with clinically significant abnormalities in 12-lead ECG results at screening, as determined by the investigator (e.g., QTcF interval (Fridericia's formula) >450 msec for males, >470 msec for females; PR interval >200 msec, etc.).
5. Subjects with systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg at screening.
6. Subjects with alanine aminotransferase (ALT) >1.5×ULN, aspartate aminotransferase (AST) >1.5×ULN, or total bilirubin (TBIL) >1×ULN at screening.
7. Pregnant or breastfeeding females.
8. Subjects who have undergone major surgery within 3 months before screening or plan to undergo surgery during the study period.
9. Subjects who are positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), or syphilis serospecific antibody (TP-Ab).
10. Subjects who are heavy smokers or have smoked an average of 5 or more cigarettes per day within 3 months before screening.
11. Subjects with difficulty in venous blood collection or who experience fainting or dizziness during blood collection.
12. Subjects who have taken any medication, including prescription drugs, over-the-counter drugs, herbal medicines, or dietary supplements, within 2 weeks or 5 half-lives (whichever is longer) before screening, and are expected to take any medication during the study period (except for the rosuvastatin treatment in Part C) (excluding treatment for adverse events).
13. Subjects with diseases or conditions that, as determined by the investigator, could significantly affect the absorption of drugs or nutrients, such as clinically significant gastrointestinal diseases (e.g., active inflammatory bowel disease) or symptoms of gastrointestinal disorders; or any condition that could affect drug absorption, such as subtotal or total gastrectomy, gastric bypass, or any bowel resection.
14. Subjects whom the investigator deems ineligible.

    Subjects with the following diseases or medical history before screening or before randomization:
15. Subjects with a history of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, or a history of hypersensitivity to drugs with a chemical structure similar to HS-10510, as determined by the investigator.
16. Subjects with a history of endocrine diseases that could significantly affect body weight, such as diabetes, Cushing's syndrome, hypothyroidism, or hyperthyroidism.
17. Subjects with a history of moderate to severe depression or a history of severe psychiatric disorders, such as schizophrenia or bipolar disorder.
18. Subjects with a history of acute or chronic hepatitis or other severe liver diseases, except for non-alcoholic fatty liver disease.
19. Subjects with a history of severe cardiovascular disease within 6 months before screening, including decompensated heart failure (NYHA class III and IV), unstable angina, stroke or transient ischemic attack, acute myocardial infarction, severe arrhythmia, or coronary artery bypass grafting or percutaneous coronary intervention.
20. Subjects with a history of or current severe infection, such as cellulitis, pneumonia, or sepsis, within 30 days before screening.
21. Subjects with a history of drug abuse or illicit drug use within 1 year before screening, or positive results on urine drug screening.
22. Subjects with a history of alcoholism or who have consumed more than 14 units of alcohol (1 unit = 285 mL of beer, 25 mL of spirits (≥35% alcohol), 150 mL of wine) in a single session within 2 weeks before screening, or positive results on alcohol breath testing at screening.
23. Subjects with a history of malignant tumors.
24. Subjects who have received or plan to receive live (attenuated) vaccines within 12 weeks before screening.
25. Subjects with concurrent cardiovascular, liver, kidney, gastrointestinal, psychiatric, neurological, hematological, or metabolic disorders.

    Subjects who have used any of the following medications or treatments before screening:
26. Subjects who have used medications that could affect cholesterol levels (e.g., statins, ezetimibe, niacin, and supplements such as ω-3 fatty acids) within 8 weeks before screening.
27. Subjects who are currently or have previously received inclisiran sodium or other investigational siRNA PCSK9 inhibitors.
28. Subjects who have received PCSK9 inhibition (approved or investigational) treatment within 12 months before screening.
29. Subjects who have received microsomal triglyceride transfer protein inhibitors (e.g., lomitapide) within 12 months before screening.
30. Subjects who have received systemic steroid therapy, immunomodulatory therapy, or chemotherapy within 3 months before screening, or who may receive these treatments during the study period.
31. Subjects who are currently receiving or have received medications known to prolong the QT interval (refer to the package insert) within 14 days before screening.

    Subjects with any of the following conditions:
32. Subjects who have participated in any drug or medical device clinical trial and received at least one treatment (including placebo) within 12 weeks before screening, or are still within 5 half-lives of the investigational drug (whichever is longer, excluding those who did not receive the investigational drug or device).
33. Subjects who are strict vegetarians or have medical dietary restrictions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events | From Screening until Follow-up Visit (7 days post-dose for all cohorts)
  The safety and tolerability of HS-10510 following oral administration of single ascending doses (Part A) and multiple ascending doses (Part B and C) will be assessed.

SECONDARY OUTCOMES:
LDL-C | SAD cohorts: Days 1,2,3,4,8 Food Effect SAD cohort: Day 1,2,3,4,8,9,10,11,15 MAD cohorts: Days1,2,3,4,7,11,15,22,26,28,31,35 Rosuvastatin MAD Cohorts: Days1,2,3,4,7,11,15,22,26,28,31,35
  The pharmacodynamics (PD) of HS-10510 by assessment of LDL-C following oral administration of single ascending doses (Part A) and multiple ascending doses (Part B and C) will be assessed.
Proprotein convertase subtilisin/kexin type 9(PCSK9) | SAD cohorts: Days 1,2,3,8 Food Effect SAD cohort: Day 1,2,3,8,9,10,15 MAD cohorts: Days 1,2,3,7,11,15,22,28,31,35 Rosuvastatin MAD Cohorts: Days 1,2,3,7,11,15,22,28,31,35
  The PD of HS-10510 by assessment of PCSK9 following oral administration of single ascending doses (Part A) and multiple ascending doses (Part B and C) will be assessed.
HS-10510 PK parameter: Maximum observed plasma concentration (Cmax) | SAD cohorts: Day 1 to Day 4 Food Effect SAD cohort: Day 1 to Day 4 and Day 8 to Day 11 MAD cohorts: Day 1 to Day 31 Rosuvastatin MAD Cohorts: Day 1 to Day 31
  To characterise the single dose and steady state PK of HS-10510 following oral administration of HS-10510.
HS-10510 PK parameter: Area under plasma concentration-time curve from zero to infinity (AUC0-inf) | SAD cohorts: Day 1 to Day 4 Food Effect SAD cohort: Day 1 to Day 4 and Day 8 to Day 11 MAD cohorts: Day 1 to Day 31 Rosuvastatin MAD Cohorts: Day 1 to Day 31
  To characterise the single dose and steady state PK of HS-10510 following oral administration of HS-10510.
HS-10510 PK parameter: Area under the plasma concentration-curve from 0 to the last quantifiable concentration (AUC0-last) | SAD cohorts: Day 1 to Day 4 Food Effect SAD cohort: Day 1 to Day 4 and Day 8 to Day 11 MAD cohorts: Day 1 to Day 31 Rosuvastatin MAD Cohorts: Day 1 to Day 31
  To characterise the single dose and steady state PK of HS-10510 following oral administration of HS-10510.
HS-10510 PK parameter: Area under the plasma concentration-curve across the dosing interval (AUC0-tau) | MAD cohorts: Day 1 to Day 31 Rosuvastatin MAD Cohorts: Day 1 to Day 31
  To characterise the steady state PK of HS-10510 following oral multiple administration of HS-10510.
HS-10510 PK parameter: Time to reach maximum observed concentration (Tmax) | SAD cohorts: Day 1 to Day 4 Food Effect SAD cohort: Day 1 to Day 4 and Day 8 to Day 11 MAD cohorts: Day 1 to Day 31 Rosuvastatin MAD Cohorts: Day 1 to Day 31
  To characterise the single dose and steady state PK of HS-10510 following oral administration of HS-10510.
HS-10510 PK parameter: Terminal elimination half-life (t½) | SAD cohorts: Day 1 to Day 4 Food Effect SAD cohort: Day 1 to Day 4 and Day 8 to Day 11 MAD cohorts: Day 1 to Day 31 Rosuvastatin MAD Cohorts: Day 1 to Day 31
  To characterise the single dose and steady state PK of HS-10510 following oral administration of HS-10510.
HS-10510 PK parameter: Apparent total body clearance (CL/F) | SAD cohorts: Day 1 to Day 4 Food Effect SAD cohort: Day 1 to Day 4 and Day 8 to Day 11 MAD cohorts: Day 1 to Day 31 Rosuvastatin MAD Cohorts: Day 1 to Day 31
  To characterise the single dose and steady state PK of HS-10510 following oral administration of HS-10510.
HS-10510 PK parameter: Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | SAD cohorts: Day 1 to Day 4 Food Effect SAD cohort: Day 1 to Day 4 and Day 8 to Day 11 MAD cohorts: Day 1 to Day 31 Rosuvastatin MAD Cohorts: Day 1 to Day 31
  To characterise the single dose and steady state PK of HS-10510 following oral administration of HS-10510.